CLINICAL TRIAL: NCT07092605
Title: Effectiveness of Microdosed GLP-1 in Improving Health, Quality of Life, and Longevity Measures: For Use in Healthy Individuals Ages 18-65 Who Seek to Improve Their Health and Longevity Through Low-dose (Microdosed) GLP1 Receptor Agonists
Brief Title: Effectiveness of Microdosed GLP-1 in Improving Health, Quality of Life, and Longevity Measures
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALRx010
Record Dates: First submitted 2024-12-18; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Longevity; Quality of Life; Mood; Inflammation; Immune Health; Pain Management; Weight Management; Alertness
Keywords: Microdosing GLP1s; Longevity; Weight Management; Quality of Life
MeSH Terms: conditions — Inflammation; Agnosia | interventions — Glucagon-Like Peptide 1; semaglutide

STUDY DESIGN:
Intervention Model Description: Single-Center, Prospective, Blinded, Randomised, Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Placebo (Placebo Comparator): Placebo administered in PCCA sub-magna compounding base only.
  Interventions: Drug: Placebo
- Sublingual GLP1 (Active Comparator): Semaglutide 1mg/1ml administered in PCCA sub-magna compounding base only.
  Interventions: Drug: GLP-1
- Subcutaneous GLP1 (Active Comparator): Semaglutide 1mg/ml x5ml
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — Sublingual GLP1 (weekly), Subcutaneous GLP1 (weekly), Sublingual Placebo (weekly) for up to 6 months.
  Other Names: Semaglutide
  Arms: Subcutaneous GLP1; Sublingual GLP1
Drug: Placebo — Sublingual Placebo (weekly) for up to 6 months
  Arms: Oral Placebo

SUMMARY:
The goal of this clinical study has two objectives. The Primary Objective is to evaluate the effectiveness of microdosed GLP-1 receptor agonists in improving measures of health, quality of life, and longevity. The Secondary Objective: To assess the impact of these therapies on weight management practices and metabolic health.

DETAILED DESCRIPTION:
Participants will be assigned to one of three groups: 1) control, 2) microdosed sublingual semaglutide, 3) microdosed subcutaneous semaglutide. At baseline and every 4 weeks thereafter, participants will be asked to complete surveys on health, wellness, mood, demographic information, and similar. Additionally, at baseline and every 12 weeks thereafter, they will be requested to complete evaluative blood work to measure CBC, CMP, and standard health biomarker panels (e.g., cholesterol, glucose, creatinine, sodium, potassium). From baseline throughout the duration of the study, participants will be given the option to share data from wearable activity and health trackers with the research team for greater accuracy in evaluating measures of activity, sleep, heart rate, and similar.

ELIGIBILITY:
Inclusion Criteria:

* New or existing AgelessRx patient
* Adults (aged 18-65)
* Any sex
* Any ethnicity
* BMI ≥ 20 kg/m^2
* Interest in taking microdoses of semaglutide for health and longevity improvement with no intent to seek weight loss improvement.

Exclusion Criteria:

* Individuals who are denied a longevity product by the AgelessRx medical team will not be asked to participate in any product specific test(s) or questionnaire(s)
* History of bariatric surgery
* Use of other weight-loss medications currently or within the past 6 months
* Contraindications to semaglutide
* Significant psychiatric illness that may affect participation
* Pregnant or breastfeeding individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported pain levels in participants microdosing GLP1s | 6 months
  Participants will complete an extensive medical questionnaire every 4 weeks over a 24-week period to monitor self-reported pain levels
Concentration of complete blood cells, as a measure of immunological health, in participants microdosing GLP1s | 6 months
  CBC panel will be analyzed every 12 weeks over a 24-week period, reported in thousands of cells per microliter with the change from baseline reported as percent deviation and compared to normalized range of healthy individuals
Concentration of basic metabolites (cholesterol, glucose, creatinine, sodium, potassium), as a measure of immunological health, in participants microdosing GLP1s | 6 months
  BMP panel will be analyzed every 12 weeks over a 24-week period, reported in mg/dL with the change from baseline reported as percent deviation and compared to a normalized range of healthy individuals
Change in mood in participants microdosing GLP1s | 6 months
  Mood will be assessed every 4 weeks over a 24-week period using the SF-36 standardized questionnaire with deviation reported as percent change from baseline
Change in heart rate variability in participants microdosing GLP1s | 6 months
  Participants will wear health devices with data monitored every 4 weeks over a 24-week period to observe change in heart rate variability, being defined as the variability of a participant's resting heart rate. Variability will be measured as an average deviation from baseline heart rate at each timepoint and reported as percent difference.
Changes in sleep patterns in participants microdosing GLP1s | 6 months
  Wearable health device data will be monitored over the 24-week period assessing REM vs non-REM sleep and reported as a ratio
Change in frequency of physical activity in participants microdosing GLP1s | 6 months
  The change in frequency of physical activity, defined as a departure from baseline in time spent performing moderate to rigorous physical exercise, will be captured via wearable health device data and will be reported as percent difference from baseline in steps taken.
Change in frequency of physical activity in participants microdosing GLP1s | 6 months
  The change in frequency of physical activity, defined as a departure from baseline in time spent performing moderate to rigorous physical exercise, will be captured via wearable health device data and will be reported as percent difference from baseline in calories burned.

SECONDARY OUTCOMES:
Variation in concentration of metabolic health biomarkers in participants microdosing GLP1s | 6 months
  Changes in HbA1c levels will be assessed every 12 weeks and reported as a percent deviation from baseline
Variation in concentration of metabolic health biomarkers in participants microdosing GLP1s | 6 months
  Changes in LDL cholesterol levels will be assessed every 12 weeks and reported as a percent deviation from baseline
Variation in concentration of metabolic health biomarkers in participants microdosing GLP1s | 6 months
  Changes in HDL cholesterol levels will be assessed every 12 weeks and reported as a percent deviation from baseline
Variation in concentration of metabolic health biomarkers in participants microdosing GLP1s | 6 months
  Changes in triglyceride levels will be assessed every 12 weeks and reported as a percent deviation from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Grieco M, Giorgi A, Gentile MC, d'Erme M, Morano S, Maras B, Filardi T. Glucagon-Like Peptide-1: A Focus on Neurodegenerative Diseases. Front Neurosci. 2019 Oct 18;13:1112. doi: 10.3389/fnins.2019.01112. eCollection 2019. PMID 31680842
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Drucker DJ. Mechanisms of Action and Therapeutic Application of Glucagon-like Peptide-1. Cell Metab. 2018 Apr 3;27(4):740-756. doi: 10.1016/j.cmet.2018.03.001. PMID 29617641
- See also: Link to AgelessRx Research page. — https://agelessrx.com/research/

DOCUMENTS (1):
  • Informed Consent Form (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT07092605/ICF_000.pdf